CLINICAL TRIAL: NCT05013229
Title: A 52 Week Study Comparing the Efficacy and Safety of Once Weekly IcoSema and Daily Insulin Glargine 100 Units/mL Combined With Insulin Aspart, Both Treatment Arms With or Without Oral Anti Diabetic Drugs, in Participants With Type 2 Diabetes Inadequately Controlled With Daily Basal Insulin. COMBINE 3
Brief Title: A Research Study to See How Well the New Weekly Medicine IcoSema, Which is a Combination of Insulin Icodec and Semaglutide, Controls Blood Sugar Level in People With Type 2 Diabetes Compared to Insulin Glargine Taken Daily With Insulin Aspart (COMBINE 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1535-4593; U1111-1260-8295 (Other: WHO); 2020-005309-18 (EudraCT Number); jRCT2051210127 (Registry Identifier: JAPIC)
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IcoSema (Experimental): Participants will receive once weekly subcutaneous (s.c) injections of IcoSema during the 52-week treatment period.
  Interventions: Drug: IcoSema
- Insuling glargine/insulin aspart (Active Comparator): Participants will receive subcutaneous (s.c) injections of insulin glargine once daily combined with 2-4 times daily injections of insulin aspart.
  Interventions: Drug: Insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: IcoSema — Participants will receive a once weekly subcutanous (s.c.) injection of IcoSema, on the same day every week for 52 weeks.
  Arms: IcoSema
Drug: Insulin glargine — Participants will receive a once daily subcutaneous (s.c.) injection of insulin glargine combined with Insulin aspart 2-4 times a day during mealtimes for 52 weeks.
  Arms: Insuling glargine/insulin aspart
Drug: insulin aspart — Participants will receive a once daily subcutaneous (s.c.) injection of insulin glargine combined with Insulin aspart 2-4 times a day during mealtimes for 52 weeks.
  Arms: Insuling glargine/insulin aspart

SUMMARY:
This study will compare the new medicine IcoSema, which is a combination of insulin icodec and semaglutide, taken once a week, to insulin glargine taken daily with insulin aspart in people with type 2 diabetes.The study will look at how well IcoSema controls blood sugar level in people with type 2 diabetes compared to insulin glargine taken with insulin aspart. Participants will either get IcoSema or insulin glargine taken with insulin aspart. Which treatment participants get is decided by chance. IcoSema is a new medicine that doctors cannot prescribe. Doctors can already prescribe insulin glargine and insulin aspart in many countries.

Participants will get IcoSema or insulin glargine together with insulin aspart. Participants must inject IcoSema once a week or inject insulin glargine once daily and insulin aspart 2-4 times a day. Participants will inject the medicines with a pen, which has a small needle, in a skin fold in the thigh, upper arm, or stomach. The study will last for about 1 year and 1 month. Participants will be asked to wear a sensor that measures participants blood sugar level all the time during an 8 week period at the beginning of the study and a 4 week period at the end of the study.

Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus 180 days or more before screening.
* HbA1c of 7.0-10.0 percentage (53.- 85.8 mmol/mol) (both inclusive) as assessed by central laboratory on the day of screening.
* Treated with once daily or twice-daily basal insulin (neutral protamine hagedorn insulin, insulin degludec, insulin detemir, insulin glargine 100 units/mL, or insulin glargine 300 units/mL) 20-80 units/day 90 days or more before screening. Short term bolus insulin treatment for a maximum of 14 days before screening is allowed, as is prior insulin treatment for gestational diabetes. The treatment can be with or without any of the following anti diabetic drugs with stable doses 90 days or more before screening:

  * Metformin
  * Sulfonylureas(a)
  * Meglitinides (glinides)(a)
  * DPP-4 inhibitors(a)
  * Sodium-glucose co-transporter 2 inhibitors
  * Alpha-glucosidase-inhibitors
  * Thiazolidinediones
  * Marketed oral combination products only including the products listed above.
* Body mass index (BMI) less than or equal to 40.0 kg/m^2.

  1. Sulfonylureas, meglitinides (glinides) and DPP-4 inhibitors must be discontinued at randomisation.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Anticipated initiation or change in concomitant medication (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid, hormones, or systemic corticosteroids).
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening.
* Any episodes of diabetic ketoacidosis within 90 days before screening. As declared by the participant or in the medical records.
* Presence or history of pancreatitis (acute or chronic) within 180 days before screening.
* Any of the following: Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days before screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Recurrent severe hypoglycaemic episodes within the last year (12 months) as judged by the investigator.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline week 0 (V2) to week 52 (V54)
  Percent-points

SECONDARY OUTCOMES:
Change in body weight | From baseline week 0 (V2) to week 52 (V54)
  Kg
Number of clinically significant hypoglycaemic episodes (level 2) (less than 3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) | From week 0 (V52) to week 52 (V54)
  Number of episodes
Time in range 3.9 - 10.0 mmol/L (70 - 180 mg/dL) using continuous glucose monitoring (CGM) system, Dexcom G6 | From week 48 (V50) to week 52 (V54)
  Percentage of readings
Time spent more than 10.0 mmol/L (180 mg/dL) using continuous glucose monitoring (CGM) system, Dexcom G6 | From week 48 (V50) to week 52 (V54)
  Percentage of readings
Time spent less than 3.0 mmol/L (54 mg/dL) using continuous glucose monitoring (CGM) system, Dexcom G6 | From week 48 (V50) to week 52 (V54)
  Percentage of readings
Change in fasting plasma glucose (FPG) | From baseline week 0 (V2) to week 52 (V54)
  mmol/L
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQs) in total treatment satisfaction | From baseline week 0 (V2) to week 52 (V54)
  Score 0-36. The higher the score the greater the satisfaction with treatment.
Number of severe hypoglycaemic episodes (level 3) | From baseline week 0 (V2) to week 57 (V56)
  Number of episodes
Number of clinically significant hypoglycaemic episodes (level 2) (less than 3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From baseline week 0 (V2) to week 57 (V56)
  Number of episodes
Weekly insulin dose (total) | From week 50 (V52) to week 52 (V54)
  Units

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (181):
- United States (66):
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - Valley Research, Fresno, California
  - Scripps Wht Diab Inst La Jolla, La Jolla, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Downtown LA Res Ctr. Inc., Los Angeles, California
  - San Diego Family Care, San Diego, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Creekside Endocrine Associates, Denver, Colorado
  - Clinical Res Of W Florida Inc, Clearwater, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Sweet Hope Research Specialty, Hialeah, Florida
  - E Coast Inst for Rsrch LLC_Jacksonville, Jacksonville, Florida
  - Northeast Res Inst. Inc., Jacksonville, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - South Broward Research LLC, Miramar, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Renstar Medical Research, Ocala, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - Endo Res Solutions Inc, Roswell, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Saltzer Medical Group Research, Nampa, Idaho
  - Endeavor Health, Skokie, Illinois
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton-O'Neil Diab & Endo Ctr, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - ActivMed Practice & Research LLC, Methuen, Massachusetts
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern NH Diabetes and Endocrinology, Nashua, New Hampshire
  - John J Shelmet, MD, Lawrenceville, New Jersey
  - Mid Hudson Med Res-New Windsor, New Windsor, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Physicians East Endocrinology, Greenville, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Central Ohio Clinical Research LLC, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - HealthStar Physicians PC, Morristown, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - PrimeCare Medical Group, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Andres Garcia-Zuniga, MD, P.A, Laredo, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Clinical Investigations Of Texas, Plano, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Amherst Family Practice P.C., Winchester, Virginia
  - Sound Medical Research, Port Orchard, Washington
  - Rainier Clin Res Ctr Inc, Renton, Washington
  - Ascension Medical Group- Germantown Clinic, Milwaukee, Wisconsin
- Czechia (13):
  - Fakultni nemocnice Plzen, Pilsen, Czech Republic
  - Ambulance Brno s.r.o., Brno
  - Fakultní nemocnice U sv. Anny v Brně, Brno
  - University Hospital U sv. Anny, Brno
  - Dum zdravi, Hodonín
  - FN Hradec Kralove, Hradec Králové
  - Klinika Dr. Pírka s.r.o., Mladá Boleslav
  - Diabet2 s.r.o., Prague
  - Diabetologická a interní ambulance Diabet2, Prague
  - III. interni klinika VFN a 1. LK UK v Praze, Prague
  - Institut klinicke a experimentalni mediciny_Praha, Prague
  - Fledip s.r.o., Prague
  - ResTrial s.r.o., Prague
- France (7):
  - Centre Hospitalier Departemental Vendee- La Roche Sur Yon, La Roche-sur-Yon
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-2, Le Creusot
  - Centre Hospitalier de Narbonne, Narbonne
  - Aphp-Hopital Lariboisiere-1, Paris
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-2, Pessac
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (7):
  - InnoDiab Forschung GmbH, Essen
  - Plassmann, Essen
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
- Hungary (6):
  - Békés Megyei Központi Kórház - dr. Réthy Pál Tagkórház, Békéscsaba
  - Clinexpert Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Szőcs Depot Egészségügyi Szolgáltató Kft., Budapest
  - Semmelweis Egyetem II. Belgyógyászati Klinika, Budapest
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Coromed SMO Kft., Pécs
- India (19):
  - Apollo Hospital, Ahmedabad, Ahmedabad, Gujarat
  - Swasthya Diabetes Care, Ahmedabad, Gujarat
  - Apollo Hospital International Ltd, Gandhinagar, Gujarat
  - Diacon Hospital Private Limited, Bangalore, Karnataka
  - Sree Gokulam Medical College & Research Foundation, Trivandrum, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - chelleram Diabetes Institute, Pune, Maharashtra
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Fortis Heart Institute and Multispeciality Hospital, Mohali, Punjab
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Nizams Institute of Medical Science, Hyderabad, Telangana
  - Yashoda hospital, Hyderabad, Telangana
  - Medanta Lucknow Hospital, Lucknow, Uttar Pradesh
  - Swasthya Diabetes Care, Ahmedabad
- Italy (7):
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, CZ
  - Pol. Uni. Campus Biomedico, Roma, RM
  - Presidio Ospedale di Cittadella Azienda ULSS 6 Euganea, Cittadella
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Ospedale Civico Partinico di Palermo, Partinico
  - IRCCS Multimedica, Sesto San Giovanni (MI)
  - Ospedale San Bassiano, Vicenza
- Japan (13):
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Asano Clinic, Kawagoe-shi, Saitama, Japan
  - Tokyo Medical Univ. Hospital_Diabetes, Metabolism and Endocrinology, Shinjuku-ku, Tokyo
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Akaicho Clinic, Chiba-shi, Chiba
  - The Institute of Medical Science, Asahi Life Foundation_Internal Medicine, Chuo-ku, Tokyo
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Minami Akatsuka Clinic, Mito-shi, Ibaraki
  - Takatsuki Red Cross Hospital_Diabetes and Endocrine Div., Osaka
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
- Malaysia (11):
  - Hospital Universiti Sains Malaysia_Kota Bharu, Kelantan, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - Hospital Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Seri Manjung, Seri Manjung, Perak
  - Hospital Ampang, Ampang, Selangor
  - University Technology MARA (UiTM) - Puncak Alam, Sungai Buloh, Selangor
  - University Technology MARA (UiTM) - Sg Buloh, Sungai Buloh, Selangor
  - Klinik Kesihatan Simpang Kuala, Alor Star
  - Miri Hospital, Miri, Sarawak
- Poland (9):
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - SNZOZ Lege Artis, Bialystok
  - Centrum Medyczne Pratia Katowice, Katowice
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - NBR Polska Tomasz Klodawski, Warsaw
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
- Slovenia (5):
  - Healthcare centre Kocevje, Kočevje
  - Healthcare Centre Koper, Koper
  - UKC Ljubljana, Endocrinology and Diabetes, Ljubljana
  - General Hospital Murska Sobota, Murska Sobota
  - General Hospital Nova Gorica_Diabetes, Nova Gorica
- South Africa (4):
  - Medi-Clinic Bloemfontein, Bloemfontein, Free State
  - Lenasia Clinical Trial Centre, Lenasia, Gauteng
  - Prof P. Joshi, Pretoria, Gauteng
  - Spoke Research Inc, Cape Town, Western Cape
- Thailand (7):
  - Maharaj Nakorn Chiang Mai Hospital_Endocrilogy, Chiang Mai, Mueang Chiang Mai District
  - King Chulalongkorn Memorial Hospital_Endocrinology, Bangkok
  - Rajavithi Hospital_Diabetes and Endocrinology, Bangkok
  - Siriraj Hospital_Dept Endocrinology, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital_Endocrilogy, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
- Turkey (Türkiye) (7):
  - Başkent Üniversitesi Adana Dr. Turgut Noyan Uygulama ve Araştırma Merkezi, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Akdeniz Üniversitesi Hastanesi- Endokrinoloji, Antalya
  - Aydın Adnan Menderes Üniversitesi Hastanesi, Aydin
  - Pamukkale Universitesi Tip Fakultesi, Denizli
  - Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi- Endokrinoloji, Istanbul
  - Dokuz Eylül Üniversitesi Araştırma Uygulama Hastanesi-Endokrinoloji, Izmir

REFERENCES:
- [Derived] Billings LK, Andreozzi F, Frederiksen M, Gourdy P, Gowda A, Ji L, Pletsch-Borba L, Suzuki R, Unnikrishnan AG, Vianna AGD. Once-weekly IcoSema versus multiple daily insulin injections in type 2 diabetes management (COMBINE 3): an open-label, multicentre, treat-to-target, non-inferiority, randomised, phase 3a trial. Lancet Diabetes Endocrinol. 2025 Jul;13(7):556-567. doi: 10.1016/S2213-8587(25)00052-X. Epub 2025 Jun 4. PMID 40482670